CLINICAL TRIAL: NCT03027843
Title: A Pilot Study of the Effect of Growth Hormone in Assisted Reproductive Technology Clinical Outcome of Poor Responder
Brief Title: The Effect of Growth Hormone in Assisted Reproductive Technology Clinical Outcome of Poor Responder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: newivf20170110
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Low Ovarian Reserve
Keywords: low ovarian reserve; growth hormone; embryo quality; live birth; clinical pregnancy
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH group (Active Comparator): patients in group mini-dose GnRH-a long protocol combine with growth hormone
  Interventions: Drug: Growth Hormone
- control group (No Intervention): patients in group mini-dose GnRH-a long protocol without growth hormone

INTERVENTIONS:
Drug: Growth Hormone — in GH group, patients have weekly injections of GH dose 14 iu, until the day of hCG.
  Other Names: somatotropin;GH;somatotrophin;somatotropic
  Arms: GH group

SUMMARY:
Assisted reproduction treatment in patients with low ovarian reserve is a big difficult clinical problem. Growth hormone (GH) is crucial in the development of follicles since preantral follicle to ovulation and can promote steroid hormones and gamete formation, increase the granular cell sensitivity,and inhibition of follicular atresia. Latest research shows that GH can improve egg quality through regulating mitochondrial function of the oocytes and increase the rate of embryo euploid. It becomes a new argument in that promotion of clinical pregnancy rate in assisted reproduction treatment. GH applied in the field of assisted reproduction 30 years experience of applicable people, but drug dosage, drug intervention time continue to explore. 2015 China assisted reproductive stimulate ovulation medicine expert consensus recommend joint GH for poor ovarian response, repeated implantation failure patients and older patients assisted fertility treatment, but not on the specific use time limit, the daily dose of drugs and curative effect. How to maximize growth hormone potential advantage in improving the egg quality bothers the clinical doctors. We had a self-controlled retrospective analyses in growth hormone application and found that the average daily injections of GH dose 2 iu for 45 days can significantly improve the embryo quality in patients with low ovarian reaction. And now long-acting recombinant human growth hormone is available, which make it convenient for patients. A forward-looking experimental is expected to answer clinical practical problems and provide proper GH regimen for low ovarian responder.

DETAILED DESCRIPTION:
This study is a pilot study to investigate the effect of growth hormone in assisted reproductive technology clinical outcome of poor responder.

Design: randomized controlled trial. Setting: Assisted reproductive technologies unit. Patients: patients diagnosed poor ovarian responder who is in accordance with the inclusion criteria, and not meet the exclusion criteria, who had repeated IVF treatment from Mar 2017 to Aug 2019.

Intervention: The comparison was made between GH group and the control group, both groups are conducted with the mini-dose GnRH-a long protocol for IVF treatment. GH group use Long-acting recombinant human growth hormone 14IU qw, until the day of hCG.

Main outcome measures: The primary outcome of the study is live birth rate. The secondary outcomes were clinical pregnancy rate, number of oocytes retrieved, fertility rate, normal fertilization rate, rate of transferable embryo and good quality embryo rate.

ELIGIBILITY:
Inclusion Criteria:

1. Women age ≥35 years and ≤40 years.
2. 2≤ AFC≤6, and AMH level ≥0.5 and≤ 1.1 ng/ml.
3. Previous failed transfer cycle ≥2
4. Didn't participate in other clinical subjects in three months.
5. Written informed consent.

Exclusion Criteria:

1. Body mass index (BMI) ≥25 kg/m2.
2. Endocrine metabolic disease, such as diabetes, insulin resistance, hyperthyroidism, Cushing's syndrome, hyperprolactinemia.
3. Hypertension (systolic blood pressure ≥140mmHg and diastolic blood pressure≥90mmHg.
4. Autoimmune diseases was definitively diagnosed, such as systemic lupus erythematosus, Sjogren's syndrome, Hashimoto's Thyroiditis, multiple sclerosis, rheumatoid arthritis, autoimmune hemolytic anemia, recurrent miscarriage.
5. Ovarian neoplasm that ≥4 cm in diameter and has no clear pathological diagnosis by surgery.
6. Complicated with adenomyosis, endometriosis confirmed by surgery, ovarian endometriosis cyst ≥2 cm by ultrasound, all kind of malignant tumors or precancerous disease.
7. Untreated hydrosalpinx.

Eliminate or falls off Criteria:

1. Withdraw drug and take appropriate treatment measures if serious adverse events happen during the trial, and subjects will be off.
2. Patients that have bad compliance.
3. Subjects are found breach the inclusion criteria, or in accordance with exclusion criteria during the test, excluded.
4. Patients request withdrawal and exit the trial because adverse events occur during the trial.
5. No record about treatment.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1-2year
  Live birth rate(%): number of live birth/ transferred cycle.Compare the live birth rate between the two group with SPSS 20.0.

SECONDARY OUTCOMES:
clinical pregnancy rate | 1-2 year
  Clinical pregnancy means pregnancy sac is seen intrauterine under ultrasound 7 weeks after embryo transferred. Clinical pregnancy rate(%): number of clinical pregnancy/transferred cycle.Compare the clinical pregnancy rate between the two group with SPSS 20.0.
number of oocytes retrieved | 1-2 year
  Compare the number of oocytes retrieved between the two group with SPSS 20.0.
fertility rate | 1-2 year
  Fertility rate(%): number of occyte fertilized/ number of oocytes retrieved. Compare the fertility rate between the two group with SPSS 20.0.
normal fertility rate | 1-2 year
  Normal fertility rate(%): number of occyte normally fertilized/ number of oocytes retrieved. Compare the normal fertility rate between the two group with SPSS 20.0.
transferable embryo rate | 1-2 year
  Cleavage embryo grades 1 or 2 with at least 5 blastomeres are considered as transferrable embryo.Transferable embryo rate(%): number of transferable embryo/number of feritilized oocytes. Compare the transferable embryo rate between the two group with SPSS 20.0.
good quality embryo rate | 1-2 year
  Cleavage embryo grades 1 or 2 with 6-10 blastomeres were considered good quality embryos. Good quality embryo rate(%): number of good quality embryo/number of feritilized oocytes.Compare the good quality embryo rate between the two group with SPSS 20.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Yang, M.D. & Ph.D., Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University

REFERENCES:
- [Derived] Sood A, Mohiyiddeen G, Ahmad G, Fitzgerald C, Watson A, Mohiyiddeen L. Growth hormone for in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD000099. doi: 10.1002/14651858.CD000099.pub4. PMID 34808697